CLINICAL TRIAL: NCT05122780
Title: PROgnostic Value of Precision Medicine in Patients With Myocardial Infarction and Non-obStructive Coronary artEries: the PROMISE Trial.
Brief Title: Prognostic Value of Precision Medicine in Patients With MINOCA (PROMISE Trial).
Acronym: PROMISE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Centro Cardiologico Monzino (Other); IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, MONTONE ROCCO ANTONIO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR-2019-12370197
Record Dates: First submitted 2021-07-23; First posted 2021-11-17 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Myocardial Infarction With Non-Obstructive Coronary Arteries
Keywords: MINOCA; coronary spasm; OCT
MeSH Terms: conditions — MINOCA; Angina Pectoris, Variant | interventions — Percutaneous Coronary Intervention; Platelet Aggregation Inhibitors; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Adrenergic beta-Antagonists; Nitrates; Anticoagulants

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 (using an online software available 24h/24h) to "precision medicine approach" vs "standard approach".
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Precision medicine approach" (Active Comparator): Comprehensive diagnostic work-up with:
  * Coronary angiography and ventriculography in all patients
  * OCT at the time of coronary angiography in the cath-lab.
  * Acetylcholine provocative test (to assess the presence of coronary vasospasm) at the time of coronary angiography in the cath-lab.
  * TE-Echo and/or CE-Echo (if distal/microvascular embolization is suspected)
  * Blood sampling for circulating biomarkers and miRNA expression profile
  * Trans-thoracic echocardiography in all patients during the index hospitalization
  * CMR in all cases during the index hospitalization.
  Targeted pharmacological treatment specific for the underlying cause:
  * DAPT ± stent implantation (if required), statins, beta-blockers, ACEi/ARB (in case of evidence of plaque rupture/erosion)
  * CCB and/or nitrates (in case of documentation of coronary vasospasm)
  * Anticoagulation (in case of coronary embolism).
  Interventions: Procedure: Coronary angiography; Diagnostic Test: OCT imaging; Procedure: Percutaneous coronary intervention (PCI):; Diagnostic Test: Acetylcholine provocative test; Diagnostic Test: TT-Echocardiography; Diagnostic Test: TE/contrast echocardiography; Diagnostic Test: Cardiac magnetic resonance; Diagnostic Test: Circulating biomarkers; Drug: Antiplatelet Drug; Drug: Statin; Drug: Beta blocker; Drug: ACEi/ARB; Drug: CCB; Drug: Nitrates; Drug: Anticoagulant
- "Standard approach" (Other): Routine diagnostic work-up with:
  * Coronary angiography and ventriculography
  * Transthoracic echocardiography in all patients during the index hospitalization
  * CMR with contrast media only if clinically indicated (i.e. to exclude myocarditis or takotsubo syndrome)
  Standard medical treatment with:
  * DAPT in all patients
  * Beta-blockers (if indicated by the clinical context, i.e. documentation of left ventricular ejection fraction <50%, tachycardia).
  * High intensity statins in all patients
  * ACEi/ARB (if clinically indicated).
  Interventions: Procedure: Coronary angiography; Diagnostic Test: TT-Echocardiography; Diagnostic Test: Cardiac magnetic resonance; Drug: Antiplatelet Drug; Drug: Statin; Drug: Beta blocker; Drug: ACEi/ARB

INTERVENTIONS:
Procedure: Coronary angiography — coronary angiography will be performed via the transradial or transfemoral approach with the use of a 6F sheath. Coronary angiography will be performed within 90 minutes from hospital admission in patients presenting with persistent ST-segment elevation, and within 48 hours in patients presenting with non-ST-segment elevation. Unfractionated heparin (initial weight-adjusted intravenous bolus of 60 IU/Kg, with repeat boluses to achieve an activated clotting time of 250 to 300 seconds) was administered in all patients. If evidence of plaque rupture
Diagnostic Test: OCT imaging — OCT imaging will be performed in the culprit artery in all patients randomized to the "precision medicine approach". A 0.014-inch guidewire will be placed distally in the target vessel and an intracoronary injection of 200 µg of nitroglycerine will be performed. Frequency domain OCT (FD-OCT) images are acquired by a commercially available system (C7 System, LightLab Imaging Inc/ St Jude Medical, Westford, MA) connected to an OCT catheter (C7 Dragonfly; LightLab Imaging Inc/ St Jude Medical, Westford, MA), which was advanced to the culprit lesion. The FD-OCT run will be performed using the integrated automated pullback device at 20 mm/s. During image acquisition, coronary blood flow will be replaced by continuous flushing of contrast media directly from the guiding catheter at a rate of 4 ml/s with a power injector in order to create a virtually blood-free environment.
  Arms: "Precision medicine approach"
Procedure: Percutaneous coronary intervention (PCI): — PCI with stent implantation will be considered in selected cases with evidences of plaque rupture
  Arms: "Precision medicine approach"
Diagnostic Test: Acetylcholine provocative test — ACh will be administered in a stepwise manner into the left coronary artery (LCA) (20-200 μg) or into the right coronary artery (RCA) (20-50 μg) over a period of 3 min with a 2-3 min interval between injections. Coronary angiography will be performed 1 min after each injection of these agents and/or when chest pain and/or ischaemic ECG shifts were observed. The decision of testing with provocative test LCA or RCA as first will be left to the discretion of the physicians; both LCA and RCA will be tested if the first test was negative. Angiographic responses during the provocative test will be assessed in multiple orthogonal views in order to detect the most severe narrowing and/or analysed by using computerized quantitative coronary angiography (QCA-CMS, Version 6.0, Medis-Software, Leiden, The Netherlands).
  Arms: "Precision medicine approach"
Diagnostic Test: TT-Echocardiography — TT-Echo will be used to calculate left and right ventricular and atrial dimensions, left and right ventricular systolic function, transmitral flow Doppler spectra, mitral and tricuspidal valve annulus tissue Doppler spectra, ejection time and stroke volume, inferior vena cava, aorta and pulmonary artery diameters and Doppler spectra, according to the recommendations of the American Society of Echocardiography.
Diagnostic Test: TE/contrast echocardiography — In patients with angiographic evidence or suspicion of distal microembolization, TE-Echo consisting of an echocardiographic probe inserted in to the oesophagus will be used to detect a hidden cardioembolic source (i.e. left atrial thrombus); in patients with suspected left ventricular source of cardioembolism, contrast echocardiography consisting of a 0.3ml solution of SONOVUE will be used.
  Arms: "Precision medicine approach"
Diagnostic Test: Cardiac magnetic resonance — CMR will be performed during hospital stay on a 1.5-T system equipped with a 32-channel cardiac coil. Patients underwent conventional CMR including cine, T2-weighted, first pass perfusion, and conventional breath-held late gadolinium enhancement (LGE).
Diagnostic Test: Circulating biomarkers — Blood sampling for circulating biomarkers and miRNA expression profile at the time or within 12 hours of coronary angiography. Blood sampling will be processed and analysed in the research laboratory of the Department of Cardiovascular Science. Biological aliquots will be preserved at XBiogem Biobank at Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome (see section 33).
  Arms: "Precision medicine approach"
Drug: Antiplatelet Drug — acetylsalicylic acid (loading dose 250mg intravenously followed by 75mg orally) + P2Y12 receptor inhibitor (i.e. Clopidogrel, 300 or 600mg loading dose orally, followed by 75 mg orally daily).
Drug: Statin — i.e. atorvastatin; dosages titrated on the patient's clinical characteristics
Drug: Beta blocker — i.e. bisoprolol; dosages titrated on blood pressure, ECG, heart rate
Drug: ACEi/ARB — i.e. ramipril; dosages titrated on blood pressure, ECG, heart rate
Drug: CCB — i.e. diltiazem; dosages titrated on blood pressure, ECG, heart rate
  Arms: "Precision medicine approach"
Drug: Nitrates — i.e. nitroglycerine; dosages titrated on blood pressure, ECG, heart rate
  Arms: "Precision medicine approach"
Drug: Anticoagulant — i.e. warfarin; the selection of the anticoagulant agent will be based on the clinical scenario, contraindications etc
  Arms: "Precision medicine approach"

SUMMARY:
The aim of our study is to evaluate if the use of a precision-medicine approach with a specific therapy tailored on the underlying pathogenic mechanism will improve the quality-of-life in MINOCA patients. The investigators further aim at investigating wherever a precision-medicine approach will improve the prognosis, healthcare related costs, and if that a different profile of plasma biomarkers and microRNAs may serve as diagnostic tools for detecting specific causes of MINOCA and to assess response to therapy. Finally, beyond its pivotal role in differential diagnosis, the investigators hypothesize that cardiac magnetic resonance (CMR) may provide a morphological and functional cardiac characterization as well as help in the prognostic stratification.

DETAILED DESCRIPTION:
PROMISE study is a randomized multicenter prospective superiority phase IV trial comparing "precision medicine approach" versus "standard of care" in improving the prognosis and/or the quality-of-life of patients presenting with MINOCA. Patients will be randomized 1:1 to "precision medicine approach" consisting of a comprehensive diagnostic work up aim at elucidating the pathophysiological mechanism of MINOCA and consequently a tailored pharmacological approach versus "standard of care" consisting of standard diagnostic algorithm and therapy for myocardial infarction.

The aim of the study is to evaluate if the use of a precision-medicine approach with a specific therapy tailored on the underlying pathogenic mechanism will improve the quality-of-life in MINOCA patients (primary objective). The investigators further aim at investigating wherever a precision-medicine approach will improve the prognosis, healthcare related costs, and if that a different profile of plasma biomarkers and microRNAs may serve as diagnostic tools for detecting specific causes of MINOCA and to assess response to therapy (secondary objectives). Finally, beyond its pivotal role in differential diagnosis, the investigators hypothesize that cardiac magnetic resonance (CMR) may provide a morphological and functional cardiac characterization as well as help in the prognostic stratification (secondary objective).

The study is a multicentre trial involving 3 centers: IRCCS Fondazione Policlinico Universitario A. Gemelli (Study Promoter), Centro Cardiologico Monzino IRCCS, IRCCS Policlinico San Donato.

It will include 180 patients aged >18 years hospitalized for MINOCA randomized 1:1 to a "precision medicine approach" consisting of a comprehensive diagnostic work-up, analysis of circulating biomarkers and micro RNA expression profile and pharmacological treatment specific for the underlying cause versus a "standard approach" consisting of routine diagnostic work-up and standard medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent to the study
* Age > 18y
* MINOCA diagnosis, defined as:

  * Acute myocardial infarction (based on Fourth Universal Definition of Myocardial Infarction Criteria):
  * Evidence of non-obstructive coronary artery disease on angiography (i.e., no coronary artery stenosis >50%) in any major epicardial vessel.
  * No specific alternate diagnosis for the clinical presentation (i.e. non-ischemic causes of myocardial injury such as sepsis, pulmonary embolism, and myocarditis).

Exclusion Criteria:

* Inability or limited capacity to give informed consent to the study
* Age < 18 y
* Pregnant and breast-feeding women or patients considering becoming pregnant during the study period will be excluded. For women of childbearing potential, the use of a highly effective contraceptive measure is required in order to be included in the study. "Highly effective contraceptive" is defined in accordance with the recommendations of the Clinical Trial Facilitation Group as a contraceptive measure with a failure rate of less than 1% per year (https://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2020_09_HMA_CTFG_Contraception_guidance_Version_1.1_updated.pdf).
* Alternate diagnosis for the clinical presentation (i.e. non-ischemic causes of myocardial injury such as sepsis, pulmonary embolism, valve disease, hypertrophic cardiomyopathy and myocarditis). Also patients presenting with Takotsubo syndrome will be excluded.
* Contraindication to contrast-enhanced CMR, eg, severe renal dysfunction (glomerular filtration rate <30 mL/min), non-CMR-compatible pacemaker or defibrillator.
* Contraindication to drugs administrated: e.g a history of hypersensitivity to drugs administrated or its excipients, significant renal and/or hepatic disease.
* Patients with comorbidities having an expected survival <1-year will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Angina status | 1-year follow-up
  Angina status will be evaluated using the single-item "angina stability scale" and the two-item "angina frequence scale" of the Seattle Angina Questionnaire (SAQ).
  Scores are calculated by summing items within a dimension and transforming it to a 0-100 scale, where 0 is the worst and 100 the best possible level of health.
  * To reduce the risk of detection and performance bias, a team of 2 cardiologists blinded to group allocation and belonging to an external cardiology unit will submit and collate the questionnaires from study participants.
eattle Angina Questionnaire (SAQ) | 1-year follow-up
  Quality of life will be evaluated using the nine-item scale of "physical limitations scale", the three-item "treatment satisfaction scale" and two-item "disease perception scale" of the Seattle Angina Questionnaire (SAQ).
  Scores are calculated by summing items within a dimension and transforming it to a 0-100 scale, where 0 is the worst and 100 the best possible level of health.
  * To reduce the risk of detection and performance bias, a team of 2 cardiologists blinded to group allocation and belonging to an external cardiology unit will submit and collate the questionnaires from study participants.

SECONDARY OUTCOMES:
Rates of major adverse cardiovascular events | 1-year follow-up
  Rates of major adverse cardiovascular events (MACE; composite of all-cause mortality; re-hospitalization for myocardial infarction, stroke or heart failure; repeated coronary angiography) will be evaluated at 1-year follow-up in MINOCA patients.
Healthcare primary related-costs | 1-year follow-up
  Healthcare primary related costs will be evaluated as mean costs (including procedures, tests, medicines).
Healthcare secondary related-costs | 1-year follow-up
  Healthcare secondary related-costs will be evaluated as mean quality adjusted life year (QALY) gained.
Healthcare secondary related-costs | 1-year follow-up
  Healthcare secondary related-costs will be evaluated as the incremental cost-effectiveness ratio (ICER) expressed as the cost per QALY.
Ability of different circulating biomarkers as diagnostic biomarker and stratification tool for specific causes of MINOCA. | during index hospitalization (at the time or within 12 hours of coronary angiography)
  Measurement of cardiac circulating biomarkers:
  -miRNAs (miR-16, miR-26a, miR-145, miR-222, miR-155-5p, miR-483-5p, miR-45): to measure miRNA reverse transcriptase polymerase chain reaction (RT-PCR) will be employed and results will be expressed in relative expression (2-ΔΔCT Method).
Ability of different circulating biomarkers as diagnostic biomarker and stratification tool for specific causes of MINOCA. | during index hospitalization (at the time or within 12 hours of coronary angiography)
  Measurement of cardiac circulating biomarkers:
  -Endothelin 1: It will be assessed through ELISA immunoassay and results will be expressed in Picograms per millilitre (pg/mL).
Ability of different circulating biomarkers as diagnostic biomarker and stratification tool for specific causes of MINOCA. | during index hospitalization (at the time or within 12 hours of coronary angiography)
  Measurement of cardiac circulating biomarkers:
  -Neuropeptide Y: It will be assessed through ELISA immunoassay and results will be expressed in Picograms per millilitre (pg/mL).
Ability of different circulating biomarkers as diagnostic biomarker and stratification tool for specific causes of MINOCA. | during index hospitalization (at the time or within 12 hours of coronary angiography)
  Measurement of cardiac circulating biomarkers:
  -soluble CD40 ligand: It will be assessed through ELISA immunoassay and results will be expressed in Picograms per millilitre (pg/mL).
Ability of CMR in evaluating different mechanisms of MINOCA and their prognostic value through morphological and functional cardiac characterization. | from day 3 to day 7 from the acute coronary event
  Morphological cardiac characterization will be assessed by measurement of left and right ventricle volumes (in ml or ml/m2).
Ability of CMR in evaluating different mechanisms of MINOCA and their prognostic value through morphological and functional cardiac characterization. | from day 3 to day 7 from the acute coronary event
  Morphological cardiac characterization will be assessed by measurement of the presence of myocardial edema using T2-weighted sequences and a 17 segments assessment model of cardiac segmentation.
Ability of CMR in evaluating different mechanisms of MINOCA and their prognostic value through morphological and functional cardiac characterization. | from day 3 to day 7 from the acute coronary event
  Morphological cardiac characterization will be assessed by measurement of the presence of defect of perfusion using first pass perfusion sequences and a 17 segments assessment model of cardiac segmentation.
Ability of CMR in evaluating different mechanisms of MINOCA and their prognostic value through morphological and functional cardiac characterization. | from day 3 to day 7 from the acute coronary event
  Morphological cardiac characterization will be assessed by measurement of the presence of fibrosis using late gadolinium enhancement sequences and a 17 segments assessment model of cardiac segmentation (estimated as LGE % of the cardiac segment involved).
Ability of CMR in evaluating different mechanisms of MINOCA and their prognostic value through morphological and functional cardiac characterization. | from day 3 to day 7 from the acute coronary event
  Morphological cardiac characterization will be assessed by measurement of the presence of myocardial infarct size (estimated as grams or % of left ventricular myocardial mass).
Ability of CMR in evaluating different mechanisms of MINOCA and their prognostic value through morphological and functional cardiac characterization. | from day 3 to day 7 from the acute coronary event
  Functional cardiac characterization will be assessed by measurement of right and left ventricles eject fraction (estimated as %).
Ability of CMR in evaluating different mechanisms of MINOCA and their prognostic value through morphological and functional cardiac characterization. | from day 3 to day 7 from the acute coronary event
  Functional cardiac characterization will be assesaed by measurement of regional kinetic abnormalities using a 17 segments assessment model of cardiac segmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Cosentino, MD, Principal Investigator — Centro Cardiologico Monzino; Riccardo Gorla, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (3):
- Italy (3):
  - Centro Cardiologico Monzino, Milan
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
  - IRCCS Policlinico San Donato, San Donato Milanese

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tamis-Holland JE, Jneid H, Reynolds HR, Agewall S, Brilakis ES, Brown TM, Lerman A, Cushman M, Kumbhani DJ, Arslanian-Engoren C, Bolger AF, Beltrame JF; American Heart Association Interventional Cardiovascular Care Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; and Council on Quality of Care and Outcomes Research. Contemporary Diagnosis and Management of Patients With Myocardial Infarction in the Absence of Obstructive Coronary Artery Disease: A Scientific Statement From the American Heart Association. Circulation. 2019 Apr 30;139(18):e891-e908. doi: 10.1161/CIR.0000000000000670. PMID 30913893
- [Background] Niccoli G, Scalone G, Crea F. Acute myocardial infarction with no obstructive coronary atherosclerosis: mechanisms and management. Eur Heart J. 2015 Feb 21;36(8):475-81. doi: 10.1093/eurheartj/ehu469. Epub 2014 Dec 18. PMID 25526726
- [Background] Del Buono MG, Montone RA, Iannaccone G, Meucci MC, Rinaldi R, D'Amario D, Niccoli G. Diagnostic work-up and therapeutic implications in MINOCA: need for a personalized approach. Future Cardiol. 2021 Jan;17(1):149-154. doi: 10.2217/fca-2020-0052. Epub 2020 Jul 6. PMID 32628045
- [Background] Safdar B, Spatz ES, Dreyer RP, Beltrame JF, Lichtman JH, Spertus JA, Reynolds HR, Geda M, Bueno H, Dziura JD, Krumholz HM, D'Onofrio G. Presentation, Clinical Profile, and Prognosis of Young Patients With Myocardial Infarction With Nonobstructive Coronary Arteries (MINOCA): Results From the VIRGO Study. J Am Heart Assoc. 2018 Jun 28;7(13):e009174. doi: 10.1161/JAHA.118.009174. PMID 29954744
- [Background] Grodzinsky A, Arnold SV, Gosch K, Spertus JA, Foody JM, Beltrame J, Maddox TM, Parashar S, Kosiborod M. Angina Frequency After Acute Myocardial Infarction In Patients Without Obstructive Coronary Artery Disease. Eur Heart J Qual Care Clin Outcomes. 2015;1(2):92-99. doi: 10.1093/ehjqcco/qcv014. Epub 2015 Jul 23. PMID 28239487
- [Background] Planer D, Mehran R, Ohman EM, White HD, Newman JD, Xu K, Stone GW. Prognosis of patients with non-ST-segment-elevation myocardial infarction and nonobstructive coronary artery disease: propensity-matched analysis from the Acute Catheterization and Urgent Intervention Triage Strategy trial. Circ Cardiovasc Interv. 2014 Jun;7(3):285-93. doi: 10.1161/CIRCINTERVENTIONS.113.000606. Epub 2014 May 20. PMID 24847016
- [Background] Jespersen L, Abildstrom SZ, Hvelplund A, Galatius S, Madsen JK, Pedersen F, Hojberg S, Prescott E. Symptoms of angina pectoris increase the probability of disability pension and premature exit from the workforce even in the absence of obstructive coronary artery disease. Eur Heart J. 2013 Nov;34(42):3294-303. doi: 10.1093/eurheartj/eht395. Epub 2013 Sep 26. PMID 24071763
- [Background] Montone RA, Niccoli G, Fracassi F, Russo M, Gurgoglione F, Camma G, Lanza GA, Crea F. Patients with acute myocardial infarction and non-obstructive coronary arteries: safety and prognostic relevance of invasive coronary provocative tests. Eur Heart J. 2018 Jan 7;39(2):91-98. doi: 10.1093/eurheartj/ehx667. PMID 29228159
- [Background] Montone RA, Niccoli G, Russo M, Giaccari M, Del Buono MG, Meucci MC, Gurgoglione F, Vergallo R, D'Amario D, Buffon A, Leone AM, Burzotta F, Aurigemma C, Trani C, Liuzzo G, Lanza GA, Crea F. Clinical, angiographic and echocardiographic correlates of epicardial and microvascular spasm in patients with myocardial ischaemia and non-obstructive coronary arteries. Clin Res Cardiol. 2020 Apr;109(4):435-443. doi: 10.1007/s00392-019-01523-w. Epub 2019 Jul 3. PMID 31270616
- [Background] Crea F, Niccoli G. Myocardial Infarction With Nonobstructive Coronary Atherosclerosis: The Need for Precision Medicine. JACC Cardiovasc Imaging. 2019 Nov;12(11 Pt 1):2222-2224. doi: 10.1016/j.jcmg.2018.09.003. Epub 2018 Oct 17. No abstract available. PMID 30343094
- [Background] Pasupathy S, Air T, Dreyer RP, Tavella R, Beltrame JF. Systematic review of patients presenting with suspected myocardial infarction and nonobstructive coronary arteries. Circulation. 2015 Mar 10;131(10):861-70. doi: 10.1161/CIRCULATIONAHA.114.011201. Epub 2015 Jan 13. PMID 25587100
- [Background] Dastidar AG, Baritussio A, De Garate E, Drobni Z, Biglino G, Singhal P, Milano EG, Angelini GD, Dorman S, Strange J, Johnson T, Bucciarelli-Ducci C. Prognostic Role of CMR and Conventional Risk Factors in Myocardial Infarction With Nonobstructed Coronary Arteries. JACC Cardiovasc Imaging. 2019 Oct;12(10):1973-1982. doi: 10.1016/j.jcmg.2018.12.023. Epub 2019 Feb 13. PMID 30772224
- [Background] Lindahl B, Baron T, Erlinge D, Hadziosmanovic N, Nordenskjold A, Gard A, Jernberg T. Medical Therapy for Secondary Prevention and Long-Term Outcome in Patients With Myocardial Infarction With Nonobstructive Coronary Artery Disease. Circulation. 2017 Apr 18;135(16):1481-1489. doi: 10.1161/CIRCULATIONAHA.116.026336. Epub 2017 Feb 8. PMID 28179398
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- [Background] Ford TJ, Stanley B, Sidik N, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, McCartney P, Corcoran D, Collison D, Rush C, Sattar N, McConnachie A, Touyz RM, Oldroyd KG, Berry C. 1-Year Outcomes of Angina Management Guided by Invasive Coronary Function Testing (CorMicA). JACC Cardiovasc Interv. 2020 Jan 13;13(1):33-45. doi: 10.1016/j.jcin.2019.11.001. Epub 2019 Nov 11. PMID 31709984
- [Background] Rosano GMC, Tousoulis D, McFadden E, Clarke J, Davies GJ, Kaski JC. Effects of neuropeptide Y on coronary artery vasomotion in patients with microvascular angina. Int J Cardiol. 2017 Jul 1;238:123-127. doi: 10.1016/j.ijcard.2017.03.024. Epub 2017 Mar 16. PMID 28476516
- [Background] Toyo-oka T, Aizawa T, Suzuki N, Hirata Y, Miyauchi T, Shin WS, Yanagisawa M, Masaki T, Sugimoto T. Increased plasma level of endothelin-1 and coronary spasm induction in patients with vasospastic angina pectoris. Circulation. 1991 Feb;83(2):476-83. doi: 10.1161/01.cir.83.2.476. PMID 1825037
- [Background] Fong SW, Few LL, See Too WC, Khoo BY, Nik Ibrahim NN, Yahaya SA, Yusof Z, Mohd Ali R, Abdul Rahman AR, Yvonne-Tee GB. Systemic and coronary levels of CRP, MPO, sCD40L and PlGF in patients with coronary artery disease. BMC Res Notes. 2015 Nov 14;8:679. doi: 10.1186/s13104-015-1677-8. PMID 26576922
- [Background] Jaguszewski M, Osipova J, Ghadri JR, Napp LC, Widera C, Franke J, Fijalkowski M, Nowak R, Fijalkowska M, Volkmann I, Katus HA, Wollert KC, Bauersachs J, Erne P, Luscher TF, Thum T, Templin C. A signature of circulating microRNAs differentiates takotsubo cardiomyopathy from acute myocardial infarction. Eur Heart J. 2014 Apr;35(15):999-1006. doi: 10.1093/eurheartj/eht392. Epub 2013 Sep 17. PMID 24046434
- [Background] Li S, Lee C, Song J, Lu C, Liu J, Cui Y, Liang H, Cao C, Zhang F, Chen H. Circulating microRNAs as potential biomarkers for coronary plaque rupture. Oncotarget. 2017 Jul 18;8(29):48145-48156. doi: 10.18632/oncotarget.18308. PMID 28624816
- [Derived] Montone RA, Cosentino N, Graziani F, Gorla R, Del Buono MG, La Vecchia G, Rinaldi R, Marenzi G, Bartorelli AL, De Marco F, Testa L, Bedogni F, Trani C, Liuzzo G, Niccoli G, Crea F. Precision medicine versus standard of care for patients with myocardial infarction with non-obstructive coronary arteries (MINOCA): rationale and design of the multicentre, randomised PROMISE trial. EuroIntervention. 2022 Dec 2;18(11):e933-e939. doi: 10.4244/EIJ-D-22-00178. PMID 35734824

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT05122780/Prot_SAP_000.pdf